CLINICAL TRIAL: NCT05978596
Title: Postural Alignment in Post-stroke Participants: Providing New Insights in the Time Course of a Misperception of Verticality and Its Characteristics
Brief Title: Time Course of a Misperception of Verticality and Its Characteristics in Post-stroke Participants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Wim Saeys, Professor Dr. Wim Saeys, Universiteit Antwerpen
Other Study IDs: CvdW
Record Dates: First submitted 2023-06-20; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Perception of verticality; Spatial neglect; Lateropulsion; Postural control; Subjective Visual Vertical; Subjective Haptic Vertical; Subjective Postural Vertical
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Little is known about the time course of verticality perception after stroke. This study aims to assess:

* The time course of verticality perception (Subjective Visual, Haptic and Postural Vertical; resp., SVV, SHV, SPV);
* The longitudinal interaction of the recovery of spatial disorders (e.g., different types of neglect, lateropulsion) with verticality perception;
* The longitudinal interaction of motor function and outcomes (such as paresis, sitting balance and standing balance) and verticality perception.

The participants will be repetitively assessed during the subacute phase post-stroke, to evaluate the time course of:

* The SVV, SHV and SPV;
* Spatial disorders (visuospatial and personal neglect, lateropulsion)
* Motor function (lower limb strength, sitting and standing balance, functionality in ADL, trunk performance)

DETAILED DESCRIPTION:
For a correct vertical alignment of the body with the gravitational vector, the patient must be able to accurately perceive verticality. Estimation of verticality is a complex process, suggested to be based on internal references derived from the integration of multisensory input (e.g. visual, vestibular and somatosensory). Due to a brain lesion, this complex process can be hampered, resulting in a deviation of the subjective vertical.

Different modalities of verticality perception can be assessed, including the Subjective Visual (SVV), Haptic (SHV) and Postural (SPV) Vertical. Previous studies reported a deviation of the subjective vertical in post-stroke patients. These deviations are associated with poorer balance performance. However, some stroke participants have more difficulties with accurately estimating a vertical position as compared to others. This increased magnitude is often seen in participants with lateropulsion or spatial neglect.

Although previous studies showed an increased deviation of the subjective vertical in post-stroke patients, little is known about the recovery of this misperception of verticality. Especially in patients with spatial disorders (e.g., lateropulsion or (different subtypes of) neglect), there is clear lack of studies assessing the longitudinal recovery of a misperception of verticality. Knowledge about the spontaneous recovery of a deviated verticality perception and its association with spatial disorders, will give insights in the role of a misperception of verticality in these disorders.

Although disturbances in perceiving verticality and decreased balance performance seems to be related, it is unclear how these disturbances exactly impacts balance and functional outcome. A longitudinal interaction between verticality perception and motor function will be evaluated.

Participants will be recruited from rehabilitation hospital Revarte (Edegem) or AZ Monica (Antwerp). Participants will be included at 3 or 5 weeks post-stroke and evaluation will take place at 3, 5, 8 and 12 weeks post-stroke. Also, in healthy participants the SVV, SHV and SPV will be evaluated to obtain normative data.

The outcome measures contain:

* Perception of verticality: SVV, SHV, SPV;
* Combination of pen-and-paper tasks and computerized tests to asses visuospatial and personal neglect;
* Clinical scales to evaluate lateropulsion;
* Clinical scales to evaluate motor function (lower limb strength, sitting balance, standing balance, functionality in ADL, trunk performance);
* Instrumented analysis to assess sitting and standing balance.

For the data-analysis Linear Mixed Models will be used, to evaluate study results and mean change over time.

ELIGIBILITY:
Inclusion Criteria:

* First-ever, MRI- or CT-confirmed, ischemic or hemorrhagic supratentorial stroke;
* Able to give written informed consent.

Exclusion Criteria:

* Bilateral lesions;
* Vestibular dysfunction, symptomatic orthostatic hypotension or other pre-existing neurological conditions that could interfere with the assessments;
* Inability to understand and follow basic verbal instructions;
* Hemianopsia or other visual field deficits (glasses or corrective lenses are allowed)

And a group of healthy controls to obtain normative data. These participants are eligible for inclusion if they are between 18 and 90 years old and do not suffer from vestibular dysfunction, symptomatic orthostatic hypotension or other neurological conditions that could interfere with the assessment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from rehabiliation hospital RevArte (Edegem) and AZ Monica (Antwerp).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective Visual Vertical constant error | Change from 3 to 5 weeks
  Reflects the difference between the perceived visual vertical and the gravitational vector, with the direction (ipsi- vs contralesional) considered.
Change in Subjective Visual Vertical constant error | Change from 5 to 8 weeks
  Reflects the difference between the perceived visual vertical and the gravitational vector, with the direction (ipsi- vs contralesional) considered.
Change in Subjective Visual Vertical constant error | Change from 8 to 12
  Reflects the difference between the perceived visual vertical and the gravitational vector, with the direction (ipsi- vs contralesional) considered.
Change in Subjective Hapic Vertical constant error | Change from 3 to 5 weeks
  Reflects the difference between the perceived haptic vertical and the gravitational vector, with the direction (ipsi- vs contralesional) considered.
Change in Subjective Hapic Vertical constant error | Change from 5 to 8 weeks
  Reflects the difference between the perceived haptic vertical and the gravitational vector, with the direction (ipsi- vs contralesional) considered.
Change in Subjective Hapic Vertical constant error | Change from 8 to 12 weeks
  Reflects the difference between the perceived haptic vertical and the gravitational vector, with the direction (ipsi- vs contralesional) considered.
Change in Subjective Postural Vertical constant error | Change from 3 to 5 weeks
  Reflects the difference between the perceived postural vertical and the gravitational vector, with the direction (ipsi- vs contralesional) considered.
Change in Subjective Postural Vertical constant error | Change from 5 to 8 weeks
  Reflects the difference between the perceived postural vertical and the gravitational vector, with the direction (ipsi- vs contralesional) considered.
Change in Subjective Postural Vertical constant error | Change from 8 to 12 weeks
  Reflects the difference between the perceived postural vertical and the gravitational vector, with the direction (ipsi- vs contralesional) considered.
Change in Subjective Visual Vertical unsigned error | Change from 3 to 5 weeks
  Reflects the difference between the perceived visual vertical and the gravitational vector, irrespective of the direction.
Change in Subjective Visual Vertical unsigned error | Change from 5 to 8 weeks
  Reflects the difference between the perceived visual vertical and the gravitational vector, irrespective of the direction.
Change in Subjective Visual Vertical unsigned error | Change from 8 to 12 weeks
  Reflects the difference between the perceived visual vertical and the gravitational vector, irrespective of the direction.
Change in Subjective Haptic Vertical unsigned error | Change from 3 to 5 weeks
  Reflects the difference between the perceived haptic vertical and the gravitational vector, irrespective of the direction.
Change in Subjective Haptic Vertical unsigned error | Change from 5 to 8 weeks
  Reflects the difference between the perceived haptic vertical and the gravitational vector, irrespective of the direction.
Change in Subjective Haptic Vertical unsigned error | Change from 8 to 12 weeks
  Reflects the difference between the perceived haptic vertical and the gravitational vector, irrespective of the direction.
Change in Subjective Postural Vertical unsigned error | Change from 3 to 5 weeks
  Reflects the difference between the perceived postural vertical and the gravitational vector, irrespective of the direction.
Change in Subjective Postural Vertical unsigned error | Change from 5 to 8 weeks
  Reflects the difference between the perceived postural vertical and the gravitational vector, irrespective of the direction.
Change in Subjective Postural Vertical unsigned error | Change from 8 to 12 weeks
  Reflects the difference between the perceived postural vertical and the gravitational vector, irrespective of the direction.
Change in Subjective Visual Vertical variability | Change from 3 to 5 weeks
  Reflects the intra-individual variability (standard deviation of the trials)
Change in Subjective Visual Vertical variability | Change from 5 to 8 weeks
  Reflects the intra-individual variability (standard deviation of the trials)
Change in Subjective Visual Vertical variability | Change from 8 to 12 weeks
  Reflects the intra-individual variability (standard deviation of the trials)
Change in Subjective Haptic Vertical variability | Change from 3 to 5 weeks
  Reflects the intra-individual variability (standard deviation of the trials)
Change in Subjective Haptic Vertical variability | Change from 5 to 8 weeks
  Reflects the intra-individual variability (standard deviation of the trials)
Change in Subjective Haptic Vertical variability | Change from 8 to 12 weeks
  Reflects the intra-individual variability (standard deviation of the trials)
Change in Subjective Postural Vertical variability | Change from 3 to 5 weeks
  Reflects the intra-individual variability (standard deviation of the trials)
Change in Subjective Postural Vertical variability | Change from 5 to 8 weeks
  Reflects the intra-individual variability (standard deviation of the trials)
Change in Subjective Postural Vertical variability | Change from 8 to 12 weeks
  Reflects the intra-individual variability (standard deviation of the trials)

SECONDARY OUTCOMES:
Trunk Control Test - item quiet siting for 30 seconds | 3, 5, 8, 12 weeks post-stroke
  Sitting, hands on lap, feet of the ground. Score from 0 to 2. Higher score means better performance.
Berg Balance Scale - item quiet standing for 2 minutes | 3, 5, 8, 12 weeks post-stroke
  Ability to stand unsupported. Score from 0 to 4. Higher score means better performance.
Motricity index - lower limbs | 3, 5, 8, 12 weeks post-stroke
  Strength of the hip flexors, knee extensors and dorsiflexors (paretic vs non paretic limb)
Line Bisection Test | 3, 5, 8, 12 weeks post-stroke
  Visuospatial neglect test
Visuospatial Search Time Test | 3, 5, 8, 12 weeks post-stroke
  Visuospatial neglect test
Fluff test | 3, 5, 8, 12 weeks post-stroke
  Personal neglect test
Tactile extinction test | 3, 5, 8, 12 weeks post-stroke
  Personal neglect test
Burke Lateropulsion Scale | 3, 5, 8, 12 weeks post-stroke
  Lateropulsion test. Score from 0-17.
Scale for Contraversive Pushing | 3, 5, 8, 12 weeks post-stroke
  Lateropulsion test. Score 0-6.
Trunk Impairment test (dynamic and coordination subscales) | 3, 5, 8, 12 weeks post-stroke
  Test to evaluate the dynamic and coordinative performance of the trunk
Weight bearing asymmetry (standing) | 3, 5, 8, 12 weeks post-stroke
  Difference in weight bearing (paretic vs non-paretic) in percentage
Broken Heart Test | 3, 5, 8, 12 weeks post-stroke
  Change in cancellation task for visuospatial neglect

CONTACTS AND LOCATIONS:
Overall Officials: Wim Saeys, Prof. Dr., Principal Investigator — Universiteit Antwerpen
Locations (2):
- Belgium (2):
  - AZ Monica, Antwerp
  - RevArte, Edegem

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Waal C, Embrechts E, Loureiro-Chaves R, Gebruers N, Truijen S, Saeys W. Lateropulsion with active pushing in stroke patients: its link with lesion location and the perception of verticality. A systematic review. Top Stroke Rehabil. 2023 Apr;30(3):281-297. doi: 10.1080/10749357.2022.2026563. Epub 2022 Feb 1. PMID 35102816
- [Background] Embrechts E, van der Waal C, Anseeuw D, van Buijnderen J, Leroij A, Lafosse C, Nijboer TC, Truijen S, Saeys W. Association between spatial neglect and impaired verticality perception after stroke: A systematic review. Ann Phys Rehabil Med. 2023 Apr;66(3):101700. doi: 10.1016/j.rehab.2022.101700. Epub 2022 Dec 1. PMID 35963568
- [Background] Perennou DA, Mazibrada G, Chauvineau V, Greenwood R, Rothwell J, Gresty MA, Bronstein AM. Lateropulsion, pushing and verticality perception in hemisphere stroke: a causal relationship? Brain. 2008 Sep;131(Pt 9):2401-13. doi: 10.1093/brain/awn170. Epub 2008 Aug 4. PMID 18678565
- [Background] Bonan IV, Leman MC, Legargasson JF, Guichard JP, Yelnik AP. Evolution of subjective visual vertical perturbation after stroke. Neurorehabil Neural Repair. 2006 Dec;20(4):484-91. doi: 10.1177/1545968306289295. PMID 17082504
- [Derived] van der Waal C, Saeys W, Truijen S, Embrechts E. Clinical Assessment of Subjective Visual and Haptic Vertical Norms in Healthy Adults. Arch Clin Neuropsychol. 2024 Nov 22;39(8):1408-1417. doi: 10.1093/arclin/acae049. PMID 38940374